CLINICAL TRIAL: NCT05360459
Title: Characterization of the Intestinal and Vaginal Microbiota in Long-term Survivors of Gynecological Cancer and Its Association With Quality of Life and Sexual Health
Brief Title: Characterization of the Intestinal and Vaginal Microbiota in Long-term Survivors of Gynecological Cancer
Status: Completed | Type: Observational
Sponsor: Maria Bailen Andrino (Other)
Collaborators: Hospital Universitario Getafe (Other)
Responsible Party: Sponsor-Investigator, Maria Bailen Andrino, Assistant Professor, Universidad Autonoma de Madrid
Organization: Universidad Autonoma de Madrid (Other)
Other Study IDs: Microbiota_ radiotherapy
Record Dates: First submitted 2022-04-05; First posted 2022-05-04 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2025-01

CONDITIONS: Genital Neoplasms, Female
Keywords: radiotherapy; microbiota
MeSH Terms: conditions — Genital Neoplasms, Female

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — vaginal swab and stool specimen
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control: Healthy postmenopausal patients (more than 12 months from the last 37 menstrual period).
- Gynecological Cancer: Women affected by cervical or endometrial cancer, in early stages, with a good prognosis for life, who have received radiotherapy with or without brachytherapy (radiotherapy) with or without concurrent chemotherapy.
  Interventions: Radiation: Exposure to radiotherapy

INTERVENTIONS:
Radiation: Exposure to radiotherapy — Characterization and quantification of intestinal and vaginal microbiota in patients affected by cervical or endometrial cancer who have received pelvic radiotherapy more than 24 months ago.
  Groups: Gynecological Cancer

SUMMARY:
The study proposes the characterization of the intestinal and vaginal microbiota in long-term radiated cervical and endometrial cancer survivors to study the association with long-term radiotherapy side effects.

DETAILED DESCRIPTION:
The human epithelial surface is colonized by a community of microorganisms, the microbiota, which disruption (dysbiosis) can impact a variety of functions, leading to inflammation, altered immunity and numerous diseases, including cancer. Pelvic cancers are among the most frequently diagnosed cancers worldwide, and pelvic radiotherapy is often an essential part of multimodal therapeutic approaches but can lead to a wide range of complications for which there is currently no treatment.

The gut microbiota is altered by radiotherapy, and a relationship between gut microbiota composition, health status, and pelvic radiotherapy has been suggested. In recent years, there has been growing evidence that radiotherapy also alters the vaginal microbiota.

The study proposes the characterization of the intestinal and vaginal microbiota in long-term radiated cervical and endometrial cancer survivors to study its association with long-term radiotherapy side effects. For this purpose, a descriptive cross-sectional study will be carried out in patients affected by cervical or endometrial cancer, in early stages, with good vital prognosis who have received radiotherapy, using healthy postmenopausal women as a control group.

If the microbiota is indeed associated with the side effects of radiotherapy, this would open the possibility of identifying predictive markers, using machine learning analysis of the patients' quality of life, and would help in the search for future therapies based on the restoration of the vaginal and intestinal microbiota. Through network analysis, it would be possible to find out which factors related to patients' diet and lifestyle could be related to dysbiosis and radiotherapy-induced adverse outcomes and poor quality of life.

ELIGIBILITY:
Inclusion Criteria:

* primary diagnosis of cervical cancer or endometrial cancer.
* who have received external radiotherapy (with or without brachytherapy, with or without concomitant chemotherapy) more than 24 months ago.
* with clinical control in the last year that evidences that they are free of disease.
* who understand Spanish and have sufficient reading level to understand the questions of the quality of life questionnaires.
* sign and date the informed consent.

Exclusion Criteria:

* Recurrent or metastatic disease.
* Treatment with antibiotics or corticosteroids (3 months prior to taking the sample).
* Extreme diets (vegetarian, vegan).
* Pregnancy or lactation.
* Documented gastrointestinal diseases (gastric or duodenal ulcers, irritable colon, ulcerative colitis, Crohn's disease).
* Alcoholism (Defined as risk consumption (20-40 gr/day in women; which would be equivalent to 2-4 gr/day)
* Oral or vaginal hormone replacement therapy.
* Spermicidal products in the last 48 hours.
* Sexual intercourse in the last 48 hours.
* Immunocompromised patients.

Control patients: healthy postmenopausal women with last menstrual period more than 12 months ago in those over 40 years of age.

Exclusion criteria (controls):

* Previous diagnosis of gynecologic or breast cancer.
* Current postmenopausal genital bleeding.
* Current vulvovaginal leucorrhea.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: - Patients of the Gynecology and Obstetrics Department of the University Hospital of Getafe.
  Getafe.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2022-05-20 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Fecal microbiota (fungal and bacterial) | Baseline
  Abundance of bacterial taxa determined by 16SRNAr gene sequencing and abundance of fungal taxa by ITS2 gene sequencing. Bacterial species will also be determined by qPCR
Vaginal microbiota (fungal and bacterial) | Baseline
  Abundance of bacterial taxa determined by 16SRNAr gene sequencing and abundance of fungal taxa by ITS2 gene sequencing. Bacterial species will also be determined by qPCR

SECONDARY OUTCOMES:
Quality of life of participants | Baseline
  Quality of life of participants with gynecological cancer determined by questionnaires: EORTC QLQ-30, EORTC QLQ-EN24 and EORTC QLQ-CX24 (European Platform of Cancer Research Quality of Life Cancer Patients questionnaire) and for healthy participants determined by MENQOL questionaire

CONTACTS AND LOCATIONS:
Overall Officials: María Bailen Andrino, PhD, Principal Investigator — Universidad Autonoma de Madrid
Locations (1):
- Hospital de Getafe, Getafe, Madrid, Spain